CLINICAL TRIAL: NCT03071666
Title: Supplementation of Vitamin B12 in Pregnancy and Postpartum on Growth and Cognitive Functioning in Early Childhood: A Randomized, Placebo Controlled Trial
Brief Title: Vitamin B12 Supplementation During Pregnancy on Cognitive Development
Acronym: VitaPreg
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other); NORCE Norwegian Research Centre AS (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CISMAC-B12; Universal Trial Number (Registry Identifier: U1111-1183-4093)
Record Dates: First submitted 2017-02-23; First posted 2017-03-07 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related; Vitamin B 12 Deficiency; Anemia
Keywords: Nepal; South Asia; Nutrition; Pregnancy; Neurodevelopment; Growth
MeSH Terms: conditions — Vitamin B 12 Deficiency; Anemia | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We will randomize women in a 1:1 ratio. The vitamin B12 supplements and the placebos will be produced specifically for this trial and be identical in taste and appearance. Each woman will be assigned a packet of medicines according to her id number. This packet will only be labeled with general information about the study and a unique id number. The list that links the id number to the randomization code will be kept with the company that produces the intervention and the placebo, and with the scientist who will generate the randomization code. This scientist will otherwise not be involved in the study. None of the investigators will have access to this list until completion of data collection and cleaning of data for the main outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B12 (Experimental): cobalamin, 50 µg per day throughout pregnancy and during the first 6 months postpartum.
  Interventions: Dietary Supplement: cobalamin
- Placebo (Placebo Comparator): Identical taste and appearance with the Experimental arm. Contains no cobalamin
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: cobalamin — Vitamin supplment tablet containing 50µg cobalamin
  Other Names: Vitamin B12
  Arms: Vitamin B12
Dietary Supplement: placebo — A tablet identical to the vitamin supplement but containing no vitamin B12
  Arms: Placebo

SUMMARY:
Scientific basis: Globally, vitamin B12 deficiency is one of the most common micronutrient deficiencies. The only relevant source of vitamin B12 is animal-source foods and poor gut function may decrease absorption. Vitamin B12 is crucial for normal cell division and differentiation, and necessary for the development and myelination of the central nervous system. Deficiency is also associated with impaired fetal and infant growth. In the proposed study we will measure the effect of daily oral vitamin B12 supplementation to pregnant women on neurodevelopment and growth of their children. We also aim to measure the impact of B12 supplementation on several other outcomes.

Study design: Individually randomized double-blind placebo controlled trial in pregnant South Asian women at risk of poor vitamin B12 status. Participants will be randomized in a 1:1 ratio.

Study participants and site: 800 pregnant women from early pregnancy. Women will be enrolled as early as possible, but no later than in week 15 of pregnancy.

Intervention: Daily administration of 50 µg of vitamin B12 from early pregnancy until 6 months after birth.

Comparator: Placebo, identical to the vitamin B12 supplements.

Outcomes: Primary: (i) neurodevelopment in children measured at 6 and 12 months of age (ii) growth in children measured by weight and length at 12 months. Secondary: (i) neurodevelopment and cognitive functioning in children at 24 months (ii) gestational age at birth, (iii) fetal and infant growth measured by weight and length at birth, after 1 month and then at 3, 6, 9, and 24 months, (iv) hemoglobin concentration in children and mothers.

Relevance for programs and public health: The results from this study can suggest new dietary guidelines for South Asian women that again can lead to improved pregnancy outcomes and neurodevelopment and cognitive functioning in South Asian children.

DETAILED DESCRIPTION:
Cobalamin (Vitamin B12) deficiency is common in many low- and middle-income countries. This is not surprising as the main source of vitamin B12 is animal source foods, which are expensive and for cultural and religious reasons often not eaten at all. We have in several studies in women and children demonstrated that poor vitamin B12 status is common in South Asia. There is also compelling evidence that vitamin B12 deficiency occurs frequently in many other settings including pregnant women .

Case studies have demonstrated harmful effects of severe vitamin B12 deficiency on the developing infant brain.The consequences of mild or subclinical vitamin deficiency are less clear but it has been shown to be associated with decreased cognitive performance in both elderly and children.

Three randomized controlled trials (RCT) have measured the effect of vitamin B12 supplementation on neurodevelopment in children: In a Norwegian trial, an intramuscular injection of B12 substantially improved motor development in six weeks old infants after one month. Another intervention study in low birth weight children in Norway recently confirmed these findings. The infants in these studies had evidence of suboptimal vitamin B12 status, but none were severely deficient. We found a beneficial effect of vitamin B12 supplementation for six months on neurodevelopment in young North Indian children.

During pregnancy, vitamin B12 is concentrated in the fetus and stored in the liver. Infants born to vitamin B12-replete mothers have stores of vitamin B12 that are adequate to sustain them for the first several months postpartum. Consequently, vitamin B12 deficiency rarely occurs before the infant is about four months old if the mother has adequate vitamin B12 status during pregnancy. However, many infants of vitamin B12-deficient breastfeeding mothers are vulnerable to B12 deficiency from an early age.

In this project we will randomise Nepalese women to receive a supplement containing 50µg cobalamin or a placebo from early pregnancy until 6 months postpartum.

Hypothesis to be tested

Principal hypothesis: Daily administration of vitamin B12 to pregnant women from early pregnancy until 6 months postpartum will:

1. Increase the scores of the Bayley Scales of Infant and Toddler Development, 3rd ed. (Bayley-III) by 0.25 SD points measured at 6 and 12 months of age.
2. Increase length for age and weight for length by 0.2 z-scores at 12 months of age.

Other hypotheses to be tested (dependent on additional funding):

1. Daily maternal administration of vitamin B12 from the start of the early pregnancy and for 6 months postpartum improves the hemoglobin concentration in the mother and infant.
2. Daily maternal administration of vitamin B12 from early pregnancy and for 6 months postpartum improves plasma vitamin B12 concentration and reduces plasma total homocysteine and methylmalonic acid concentration in the mother and infant.
3. Daily maternal administration of vitamin B12 from early pregnancy and for 6 months postpartum improves insulin sensitivity in the offspring.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mother in early pregnancy and not later than 15 weeks of pregnancy.
* Current resident and plan to reside in Bhaktapur district for at least the next 2 years.
* Age of mother between 18 and 40 years.
* Consent to participate in the study.

Exclusion Criteria:

* Taking or plan to take dietary or multivitamin supplements containing vitamin B12.
* Known case of chronic disease like asthma, tuberculosis, diabetes, hypertension, hypo or hyperthyroidism or others
* Known case of current high risk pregnancy
* Severe anemia (hemoglobin concentration <7 g/dL).
* Where the study doctor finds it necessary to treat the woman with vitamin B12 or vitamin B12 containing supplements

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study target pregnant women.
Enrollment: 800 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Length | 12 months of age
  Length measured in centimeters and expressed as z-scores
Neurodevelopment | measured 6 and 12 months of age
  Cognitive composite score of the Bayley Scales of Infant and Toddler Development, 3rd ed. (Bayley-III)

SECONDARY OUTCOMES:
Child hemoglobin concentration | measured 6 and 12 months of age
  Hemoglobin measured by hemocue in full blood
Child development ASQ | 12 first months of life
  Total and subscale scores of the Ages and Stages Questionnaire - 3rd ed.
Child development Bayley | measured 6 and 12 months of age
  Subscale scores of the Bayley Scales of Infant and Toddler Development, 3rd ed. (Bayley-III)
Heart rate variability | 12 first months of life
  Heart rate variability or vagal tone
Sleep and activity | 12 first months of life
  Sleep and activity measured by Actigraph (Actiwatch)
The Infant Motor Performance | 2 months after birth
  Screening tool to assess motor development
Still births | Birth.
  Number of still births
Maternal hemoglobin concentration | at end of pregnancy and 6 and 12 months post party.
  Hemoglobin measured by hemocue in full blood
Number of complicated births | Birth.
  Number of births that were complicated
Children born at small for gestational age | Birth
  Number of children born at small for gestational age
Birth weight | Birth
  weight in g
Low birth weight | Birth
  Birthweight < 2,500 g
Very low birth weight | Birth
  Birthweight < 2,000 g
High birth weight | Birth
  Birthweight > 4,000 g

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Strand, MD/PhD, Principal Investigator — University of Bergen; Laxman Shestha, MD, Principal Investigator — Tribhuvan University; Ram K Chandyo, MD/PhD, Principal Investigator — Kathmandu University
Locations (1):
- Manjeswori Ulak, Bhaktapur, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with other researchers upon request after completion of the study (data collection) and after publication of the main outcomes. And if the ethical review boards approve the use of the data for other purposes that what is described in the proposal.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Background] Allen LH. Causes of vitamin B12 and folate deficiency. Food Nutr Bull. 2008 Jun;29(2 Suppl):S20-34; discussion S35-7. doi: 10.1177/15648265080292S105. PMID 18709879
- [Background] Samuel TM, Duggan C, Thomas T, Bosch R, Rajendran R, Virtanen SM, Srinivasan K, Kurpad AV. Vitamin B(12) intake and status in early pregnancy among urban South Indian women. Ann Nutr Metab. 2013;62(2):113-22. doi: 10.1159/000345589. Epub 2013 Jan 22. PMID 23344013
- [Background] Taneja S, Bhandari N, Strand TA, Sommerfelt H, Refsum H, Ueland PM, Schneede J, Bahl R, Bhan MK. Cobalamin and folate status in infants and young children in a low-to-middle income community in India. Am J Clin Nutr. 2007 Nov;86(5):1302-9. doi: 10.1093/ajcn/86.5.1302. PMID 17991639
- [Background] Ulak M, Chandyo RK, Adhikari RK, Sharma PR, Sommerfelt H, Refsum H, Strand TA. Cobalamin and folate status in 6 to 35 months old children presenting with acute diarrhea in Bhaktapur, Nepal. PLoS One. 2014 Mar 3;9(3):e90079. doi: 10.1371/journal.pone.0090079. eCollection 2014. PMID 24594935
- [Background] Dror DK, Allen LH. Effect of vitamin B12 deficiency on neurodevelopment in infants: current knowledge and possible mechanisms. Nutr Rev. 2008 May;66(5):250-5. doi: 10.1111/j.1753-4887.2008.00031.x. PMID 18454811
- [Background] Strand TA, Taneja S, Ueland PM, Refsum H, Bahl R, Schneede J, Sommerfelt H, Bhandari N. Cobalamin and folate status predicts mental development scores in North Indian children 12-18 mo of age. Am J Clin Nutr. 2013 Feb;97(2):310-7. doi: 10.3945/ajcn.111.032268. Epub 2013 Jan 2. PMID 23283502
- [Background] Torsvik I, Ueland PM, Markestad T, Bjorke-Monsen AL. Cobalamin supplementation improves motor development and regurgitations in infants: results from a randomized intervention study. Am J Clin Nutr. 2013 Nov;98(5):1233-40. doi: 10.3945/ajcn.113.061549. Epub 2013 Sep 11. PMID 24025626
- [Background] Kvestad I, Taneja S, Kumar T, Hysing M, Refsum H, Yajnik CS, Bhandari N, Strand TA; Folate and Vitamin B12 Study Group. Vitamin B12 and Folic Acid Improve Gross Motor and Problem-Solving Skills in Young North Indian Children: A Randomized Placebo-Controlled Trial. PLoS One. 2015 Jun 22;10(6):e0129915. doi: 10.1371/journal.pone.0129915. eCollection 2015. PMID 26098427
- [Background] Duggan C, Srinivasan K, Thomas T, Samuel T, Rajendran R, Muthayya S, Finkelstein JL, Lukose A, Fawzi W, Allen LH, Bosch RJ, Kurpad AV. Vitamin B-12 supplementation during pregnancy and early lactation increases maternal, breast milk, and infant measures of vitamin B-12 status. J Nutr. 2014 May;144(5):758-64. doi: 10.3945/jn.113.187278. Epub 2014 Mar 5. PMID 24598885
- [Background] Taneja S, Strand TA, Kumar T, Mahesh M, Mohan S, Manger MS, Refsum H, Yajnik CS, Bhandari N. Folic acid and vitamin B-12 supplementation and common infections in 6-30-mo-old children in India: a randomized placebo-controlled trial. Am J Clin Nutr. 2013 Sep;98(3):731-7. doi: 10.3945/ajcn.113.059592. Epub 2013 Jul 31. PMID 23902779
- [Background] Strand TA, Taneja S, Kumar T, Manger MS, Refsum H, Yajnik CS, Bhandari N. Vitamin B-12, folic acid, and growth in 6- to 30-month-old children: a randomized controlled trial. Pediatrics. 2015 Apr;135(4):e918-26. doi: 10.1542/peds.2014-1848. PMID 25802345
- [Background] Kumar T, Taneja S, Yajnik CS, Bhandari N, Strand TA; Study Group. Prevalence and predictors of anemia in a population of North Indian children. Nutrition. 2014 May;30(5):531-7. doi: 10.1016/j.nut.2013.09.015. Epub 2013 Oct 15. PMID 24560137
- [Background] Yajnik CS, Deshpande SS, Jackson AA, Refsum H, Rao S, Fisher DJ, Bhat DS, Naik SS, Coyaji KJ, Joglekar CV, Joshi N, Lubree HG, Deshpande VU, Rege SS, Fall CH. Vitamin B12 and folate concentrations during pregnancy and insulin resistance in the offspring: the Pune Maternal Nutrition Study. Diabetologia. 2008 Jan;51(1):29-38. doi: 10.1007/s00125-007-0793-y. Epub 2007 Sep 13. PMID 17851649
- [Derived] Strand TA, Averina M, Bakken KS, Basnet S, Bottcher Y, Huber S, Hysing M, Kvestad I, Luders T, McCann A, Pokhrel D, Ranjitkar S, Sharma AK, Shrestha M, Ulak M, Chandyo RK. Early life exposures, neurodevelopment, and health outcomes - a study protocol for a birth cohort study in Nepal. JMIR Res Protoc. 2026 Jan 5. doi: 10.2196/78593. Online ahead of print. PMID 41493372
- [Derived] Kvestad I, Ulak M, McCann A, Chandyo RK, Hysing M, Schwinger C, Ranjitkar S, Ueland PM, Basnet S, Strand TA. The Effect of Vitamin B-12 Supplementation During Pregnancy on Early Motor Performance: Secondary Analyses From a Double-Blinded Randomized Controlled Trial. J Nutr. 2025 Dec 27:101305. doi: 10.1016/j.tjnut.2025.101305. Online ahead of print. PMID 41461260
- [Derived] Chandyo RK, Kvestad I, Ulak M, Ranjitkar S, Hysing M, Shrestha M, Schwinger C, McCann A, Ueland PM, Basnet S, Shrestha L, Strand TA. The effect of vitamin B12 supplementation during pregnancy on infant growth and development in Nepal: a community-based, double-blind, randomised, placebo-controlled trial. Lancet. 2023 May 6;401(10387):1508-1517. doi: 10.1016/S0140-6736(23)00346-X. Epub 2023 Apr 6. PMID 37031691
- [Derived] Chandyo RK, Ulak M, Kvestad I, Shrestha M, Ranjitkar S, Basnet S, Hysing M, Shrestha L, Strand TA. The effects of vitamin B12 supplementation in pregnancy and postpartum on growth and neurodevelopment in early childhood: Study Protocol for a Randomized Placebo Controlled Trial. BMJ Open. 2017 Aug 29;7(8):e016434. doi: 10.1136/bmjopen-2017-016434. PMID 28851784
- See also: Centre for Intervention Science in Maternal and Child health — http://cismac.org

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT03071666/SAP_000.pdf